CLINICAL TRIAL: NCT00004326
Title: Hippocampal Complex Volume and Memory Dysfunction in Cushing's Syndrome
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Other Study IDs: 199/11872; UMMC-1043
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's syndrome; endocrine disorders; rare disease
MeSH Terms: conditions — Cushing Syndrome; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES: I. Evaluate whether chronic hypercortisolemia is specifically toxic to hippocampal cells and causes structural reduction of hippocampal volume in patients with Cushing's syndrome.

II. Determine whether reduced hippocampal volume is associated with specific memory dysfunction.

III. Examine the relationships of adrenal androgen to hippocampal volume and memory dysfunction.

IV. Examine the reversibility of hippocampal structural changes and cognitive dysfunction after cortisol levels are normalized.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo a psychiatric evaluation for mood and cognition during confirmation of diagnosis. Neuropsychologic exams include pencil and paper test and a cognitive assessment.

Endocrine studies include dexamethasone and corticotropin-releasing hormone stimulation tests. The hippocampal complex volume is assessed with coronal magnetic resonance imaging.

There is a follow-up 1 year after the initiation of treatment.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Adults and teenagers with untreated, spontaneous active Cushing's syndrome
* Diagnosis verified at the University of Michigan Medical Center, including the following: Excessive cortisol secretion measured by urinary-free cortisol, cortisol secretion rate, and plasma cortisol level
* Lack of normal circadian cortisol secretion and failure to suppress following 2 mg of dexamethasone

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 1994-08

CONTACTS AND LOCATIONS:
Overall Officials: Monica N. Starkman, Study Chair — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States